CLINICAL TRIAL: NCT02394535
Title: Combining Abraxane With Capecitabine and Radiation Therapy for Consolidation of Treatment Following Induction Chemotherapy for Locally Advanced Pancreatic Cancer
Brief Title: Nab-Paclitaxel, Capecitabine, and Radiation Therapy Following Induction Chemotherapy in Treating Patients With Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0469; NCI-2015-00516 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0469 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Borderline Resectable Pancreatic Adenocarcinoma; Locally Advanced Pancreatic Adenocarcinoma; Pancreatic Adenocarcinoma; Stage II Pancreatic Cancer AJCC v6 and v7; Stage IIA Pancreatic Cancer AJCC v6 and v7; Stage IIB Pancreatic Cancer AJCC v6 and v7; Stage III Pancreatic Cancer AJCC v6 and v7
MeSH Terms: interventions — Capecitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, radiation therapy) (Experimental): Patients receive nab-paclitaxel IV over 30 minutes on days 1, 8, 15, 22, and 29 and capecitabine PO BID on days 1-5 (Monday-Friday). Patients also undergo radiation therapy QD on days 1-5 (Monday-Friday). Treatment continues for 51/2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine; Other: Laboratory Biomarker Analysis; Drug: Nab-paclitaxel; Other: Questionnaire Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; paclitaxel albumin-stabilized nanoparticle formulation; Protein-bound Paclitaxel
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation

SUMMARY:
This phase I trial studies the side effects and best dose of nab-paclitaxel when given together with capecitabine and radiation therapy following first treatment with chemotherapy (induction therapy) in treating patients with pancreatic cancer that is not spread to tissue far away but is not operable due to abutment or encasement of blood vessels nearby (locally advanced). Drugs used in chemotherapy, such as nab-paclitaxel and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Giving nab-paclitaxel, capecitabine, and radiation therapy together may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of combining nab-paclitaxel (abraxane) with capecitabine and radiation (radiation therapy) for consolidating treatment after induction chemotherapy for locally advanced pancreatic cancer.

SECONDARY OBJECTIVES:

I. To evaluate whether combining abraxane with capecitabine and radiation for consolidating treatment after induction chemotherapy for locally advanced pancreatic cancer increases overall survival.

II. To analyze fine needle aspiration (FNA) or core needle biopsy samples for mothers against decapentaplegic homolog 4 (SMAD4) by immunocytochemistry.

III. To evaluate plasma cytokines levels, circulating tumor cells before, during and after therapy.

IV. To evaluate patient-reported symptoms using the MD Anderson Symptom Inventory Gastrointestinal Cancer Module (MDASI-GI).

V. To evaluate response rate in patients treated at the maximum tolerated dose (MTD).

OUTLINE: This is a dose-escalation study of nab-paclitaxel.

Patients receive nab-paclitaxel intravenously (IV) over 30 minutes on days 1, 8, 15, 22, and 29 and capecitabine orally (PO) twice daily (BID) on days 1-5 (Monday-Friday). Patients also undergo radiation therapy once daily (QD) on days 1-5 (Monday-Friday). Treatment continues for 5 1/2 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4-6 weeks and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Cytologic or histologic proof of adenocarcinoma of the pancreas; patients can have tumor which is locally advanced or borderline resectable; unequivocal metastases and islet cell tumors are not eligible
* All patients must be staged with a physical exam, computed tomography (CT) of the chest and contrast-enhanced helical thin-cut abdominal CT; unresectability is defined by CT criteria:

  * Evidence of tumor extension to the celiac axis or superior mesenteric (SM) artery, or
  * Evidence on either CT or angiogram of occlusion of the SM vein or SM/portal vein confluence
* Patients must have received prior induction chemotherapy for at least 2 months and up to 8 months; at least three weeks should have elapsed after the last chemotherapy
* Platelets > 100,000 cells/mm^3
* Hemoglobin > 9.0 g/dL
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3
* Bilirubin =< 1.5 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x upper limit of normal
* Alkaline phosphatase < 2.5 x upper limit of normal
* Blood urea nitrogen (BUN) < 30 mg/dL
* Creatinine =< 1.5 mg/dL or creatinine clearance > 30 ml/min (estimated as calculated with Cockcroft-Gault equation)
* Patients must have signed informed consent indicating that they are aware of the investigational nature of the study, and are aware that participation is voluntary
* Patients must have < grade 2 pre-existing peripheral neuropathy (per Common Terminology Criteria for Adverse Events [CTCAE])
* Patients must have recovery from other clinically significant, non-hematologic toxicities to =< grade 2
* Women of childbearing potential and sexually active males must use an effective contraception method during treatment and for three months after completing treatment
* Negative serum or urine beta-human chorionic gonadotropin (hCG) pregnancy test at screening for female patients of childbearing potential

Exclusion Criteria:

* Prior abdominal radiotherapy
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in any other experimental drug study
* Prior severe infusion reaction (bronchospasm, stridor, urticaria and/or hypotension) to a taxane therapy
* Prior unanticipated severe reaction to fluoropyrimidine therapy or known hypersensitivity to 5-fluorouracil
* Prior history of cancer within the last three years except for basal cell carcinoma of the skin or carcinoma in situ of the cervix; patients with previous malignancies but without evidence of disease for 3 years will be allowed to enter the trial
* Pregnant or lactating women; women of childbearing potential with either a positive or no pregnancy test at baseline; women/men of childbearing potential not using a reliable contraceptive method (oral contraceptive, other hormonal contraceptive, intrauterine device, diaphragm or condom); (postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential); patients must agree to continue contraception for 30 days from the date of the last study drug administration
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome or inability to swallow
* Known, existing uncontrolled coagulopathy, international normalized ratio (INR) > 1.5
* Patients on Coumadin must be changed to Lovenox at least 1 week prior to starting capecitabine; low dose (1 mg) Coumadin is allowed; intravenous and low-molecular weight heparin are permitted
* Patients taking sorivudine or brivudine must be off of these drugs for 4 weeks prior to starting capecitabine; patients taking cimetidine must have this drug discontinued; ranitidine or a drug from another anti-ulcer class can be substituted for cimetidine if necessary; if patient is currently receiving allopurinol, must discuss with principal investigator (PI) to see of another agent may substitute for it
* Inability to comply with study and/or follow-up procedures
* History of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis or pulmonary hypersensitivity pneumonitis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose defined as the highest dose level in which 6 patients have been treated with at most 1 instance of dose limiting toxicity (DLT) according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 4-6 weeks
  Descriptive statistics will be used to summarize will be used to summarize patient demographic and clinical characteristics as well as the incidence of DLTs at each dose level.

SECONDARY OUTCOMES:
Overall survival | Up to 4 years
  The probabilities of overall survival will be estimated using the method of Kaplan and Meier.
Response rate | Up to 4 years
  The response rate for patients treated at the maximum tolerated dose will be estimated, along with the exact 95% confidence interval.
Changes in MD Anderson Symptom Inventory Gastrointestinal Cancer Module (MDASI) | Baseline to up to 4 years
  Descriptive statistics will be used to summarize patients' MDASI data. Paired t-test or Wilcoxon sign rank test will be used to assess the change of MDASI from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene J Koay, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson in Katy, Houston, Texas
  - MD Anderson Cancer Center - League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - MD Anderson in The Woodlands, The Woodlands, Texas

REFERENCES:
- [Derived] Koay EJ, Zaid M, Aliru M, Bagereka P, Van Wieren A, Rodriguez MJ, Jacobson G, Wolff RA, Overman M, Varadhachary G, Pant S, Wang H, Tzeng CW, Ikoma N, Kim M, Lee JE, Katz MH, Tamm E, Bhosale P, Taniguchi CM, Holliday EB, Smith GL, Ludmir EB, Minsky BD, Crane CH, Koong AC, Das P, Wang X, Javle M, Krishnan S. Nab-Paclitaxel, Capecitabine, and Radiation Therapy After Induction Chemotherapy in Treating Patients With Locally Advanced and Borderline Resectable Pancreatic Cancer: Phase 1 Trial and Imaging-based Biomarker Validation. Int J Radiat Oncol Biol Phys. 2022 Nov 1;114(3):444-453. doi: 10.1016/j.ijrobp.2022.06.089. Epub 2022 Jul 18. PMID 35863672
- See also: MD Anderson Cancer Center — http://www.mdanderson.org